CLINICAL TRIAL: NCT04239664
Title: Acceptance Based Telephone Support Around the Time of Transition to Secondary Progressive Multiple Sclerosis: A Feasibility Randomised Controlled Trial
Brief Title: Acceptance Based Telephone Support When Transitioning to SPMS
Acronym: AT-SPMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19019
Record Dates: First submitted 2019-12-06; First posted 2020-01-27 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-01

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance Based Telephone Support (ABS+UC) (Experimental): One face-to-face session to be informed of the group they have been randomised into and Acceptance Based Support, followed by five 30-minute telephone sessions of Acceptance Based Support. Usual care continues as normal.
  Interventions: Other: Acceptance Based Telephone Support (ABS+UC)
- Usual Care (Control Group) (UC) (No Intervention): One face to face session to be informed of the group they have been randomised into and encouraged to ask any questions, and will be informed they will be contacted again in 8 weeks. Usual care continues as normal.

INTERVENTIONS:
Other: Acceptance Based Telephone Support (ABS+UC) — Support based on Acceptance and Committment Therapy (Hayes, 1999)
  Arms: Acceptance Based Telephone Support (ABS+UC)

SUMMARY:
What is the purpose of the study?

People with Multiple Sclerosis often say that they feel less support is available after they are diagnosed with Secondary Progressive Multiple Sclerosis, compared to before they received this diagnosis. People sometimes experience a lessening of support, despite their physical symptoms becoming more severe from both professionals and those in their personal lives. The purpose of this study is to see whether providing some telephone support to those who have recently received a diagnosis of Secondary Progressive Multiple Sclerosis is experienced as helpful and is possible to do practically. This study will help the investigators understand which type of support may be helpful for patients in the future and may pave the way for larger studies and changes to NHS provision.

Who is it for?

Participants will be those who have transitioned recently (within the last year) to Secondary Progressive Multiple Sclerosis. The investigators are inviting 40 participants to take part.

What will happen to participants if they take part?

Participants will be asked by their Neurologist or MS Nurse to take part in the study and will provide written consent to be contacted, which will be stored by the research team. Their details will be passed to the study team at the University of Nottingham, who will telephone the participant within a week to tell them a bit more about the study and ensure they are suitable for the study by asking them some questions. Following this, the participant will be sent some paper or online questionnaires to complete and return. After this, the researcher will visit the participant face to face to introduce themselves and answer any questions they may have. They will also tell the participants what "group" they have been randomly put into. There are two groups.

Those in the first group would be asked to commit to receiving a 30 minute support phonecall each week for five weeks in addition to any usual care, and the second group will receive their usual NHS care. The support phonecalls will draw from techniques used in a type of psychological therapy (acceptance and commitment therapy). All the phonecalls can be done whilst the participant is at home or in a quiet place of their choosing. After this, both groups will fill in some more paper questionnaires eight and twelve weeks after the start of the study. The investigators expect that participants will be involved in the study for around 4 months.

After the study, participants will also have the opportunity to feedback how they experienced being a participant in the study. Their responses will help the researchers understand their experience, and help them use this to think about how to adapt similar studies in the future.

DETAILED DESCRIPTION:
Brief Summary

Introduction

People with Multiple Sclerosis often say that they feel less support is available after they are diagnosed with Secondary Progressive Multiple Sclerosis, compared to before they received this diagnosis. People sometimes experience a lessening of support, despite their physical symptoms becoming more severe from both professionals and those in their personal lives. The purpose of this study is to see whether providing some telephone support to those who have recently received a diagnosis of Secondary Progressive Multiple Sclerosis is experienced as helpful and is possible to do practically. This study will help the investigators understand which type of support may be helpful for patients in the future and may pave the way for larger studies and changes to NHS provision.

Objectives

To assess the feasibility of providing a low-resource acceptance-based telephone support intervention around the time of transition to Secondary Progressive Multiple Sclerosis

Trial Configuration

A single centre, mixed-methods feasibility randomised controlled trial (RCT), comparing two groups: (1) Acceptance Based Support + usual care; (2) usual care.

Setting Secondary care. Single centre: Nottingham Hospital and community

Sample size estimate N maximum: 40 people with Secondary Progressive Multiple Sclerosis (SPMS) (20 participants per group)

In addition to this, the investigators aim to recruit 12 of the participants for the nested qualitative study.

Number of participants

The proposed number of participants for the study will be: 40 The proposed number of participants for the interviews will be: 12

Description of interventions

Acceptance Based Telephone Support (ABS+UC): One face-to-face session to be informed of the group they have been randomised into and Acceptance Based Support, followed by five 30-minute telephone sessions of Acceptance Based Support. Usual care continues as normal.

Usual Care (Control Group) (UC): One face to face session to be informed of the group they have been randomised into and encouraged to ask any questions, and will be informed they will be contacted again in 8 weeks. Usual care continues as normal.

Duration of study

The study will take place over an 8-month period from September 2019 - April 2020.

Participation in the study will take each participant 4 months.

Data Collection: September 2019-February 2020 Analysis: February 2020-April 2020

Randomisation and blinding

Once the decision to include a person with MS is made, they will be randomised to one of two groups in a ratio of 1:1: (1) ABS+UC or (2) UC. Block randomisation of 2, 4, 6 and 8 will be used to ensure parity between groups, and randomly selected block sizes will be used. Randomisation will be conducted using an online sealed envelope service (www.sealedenvelope.com), to generate a priori the random allocation sequence. Due to the nature of the intervention, the pwMS and CM delivering the treatment cannot be blinded to group allocation, but outcome assessors will be blinded. Analysis will also be undertaken blinded to group allocation.

Statistical methods

Quantitative analysis: As a feasibility trial, the main analysis will be descriptive and focus on confidence interval estimation and not formal hypothesis testing. Descriptive statistics will be used to describe outcomes and to inform power and sample size calculations for a future trial. Rates of consent, recruitment and follow-up by randomised groups will be reported. Based on the characteristics of the data, appropriate parametric and non-parametric statistics will be used to describe trends.

Qualitative analysis: Framework approach

Extended Summary

INTRODUCTION

Multiple Sclerosis (MS) is the most common neurological condition affecting young adults. For the majority people with MS (pwMS), it presents initially as a series of relapses, each followed by a period of recovery. When there is a lack of disease progression between these relapses; this is referred to as Relapsing-Remitting MS (RRMS). For many of those with RRMS, this develops into a progressive disorder with an absence of relapse then recovery, but more typically a gradual decline in function. This is called Secondary Progressive Multiple Sclerosis (SPMS), and is defined by progressive accumulation of disability after an initial RRMS course; which may or may not contain sharp episodes of decline during progression. This progression from RRMS to SPMS happens within 15 years of initial diagnosis in 50% of cases and takes a median of 20 years.

There is a significant clinical challenge for health professionals in objectively identifying the transition from RRMS to SPMS in individuals due to subtle changes in symptoms, and receiving a new diagnosis can take an average of almost three years after onset of progressive symptoms. From a psychosocial perspective, the transition from RRMS to SPMS is a very difficult time for pwMS fraught with uncertainty. Clinicians describe the impact on pwMS as receiving an SPMS diagnosis as having a similar effect of receiving the initial diagnosis. Some of the challenges faced during this period are an adjustment towards unremitting symptoms, a withdrawal of previous disease-modifying treatments, and ever greater activity limitations.

It has been argued that transition to SPMS is a 'fear-point' of the disease, a crucial and vulnerable time where ineffective support and insufficient communication can lead to patients feeling 'devastated and demoralised', but where well placed 'supportive, encouraging and compassionate' communications can be effective in addressing the attitudinal and psychological aspects of the patient, and act as a 'buffer' for the emotional morbidity associated with MS. In this vulnerable time, communication with pwMS ought to be considered foundational to effective MS care, and that 'doing something rather than nothing can be extremely important'. Loss of social support has been shown to be associated with depression, in a population which is already susceptible to mood disorders due to being a neurological and chronic condition.

The most consistent finding of a systematic review of the psychological factors that affect adjustment in pwMS found that perceived stress and certain emotion focussed coping strategies were related to worse adjustment. A strong predictor of health status in MS is self-efficacy, which may represent an important source of coping with the burdens of MS.

Exploring the way in which pwMS regulate and cope with emotion therefore is a key consideration. CBT states that modifying dysfunctional cognitions that contribute to psychological distress is a cornerstone of the therapy process, and a central mediator of therapeutic outcome. In contrast, ACT states that facilitating acceptance of emotional and cognitive content is a central part of the therapeutic process. These differences can be summarised as cognitive "reappraisal" in CBT or "acceptance" in ACT ways of regulating emotion. These ways of regulating emotion have been compared in a study into the effects of anxious arousal, which found that both cognitive reappraisal and acceptance strategies were more effective than suppression for moderating physiological sensations, with the cognitive reappraisal generally the most adaptive strategy in terms of reducing anxiety response.

In an NHS currently plagued by understaffed services, a sufficiently effective, low resource psychological telephone support, which seeks to improve self-efficacy and techniques of emotional coping is needed for those with SPMS. This study will assess the feasibility of such an intervention, which is likely to appeal to pwMS, overworked healthcare staff, and funders if it leads to a reduction in SPMS patients use of other services. The content of this telephone support may benefit from a more acceptance-based regulation of emotion considering the client group: in secondary progressive multiple sclerosis, negative illness beliefs and distress may be entirely logical due to the debilitating nature of their condition which may make CBT "reappraisal" unrealistic. For this reason, several previous authors have argued ACT has utility over existing therapeutic models in long term conditions and due to its growing evidence base and strong face validity, is being widely adopted by health professionals working with long term conditions.

PURPOSE

As the AT-SPMS intervention is a 'complex intervention' (based on Medical Research Council [MRC] definition); the investigators aim to evaluate the key feasibility parameters before proceeding to a randomised controlled trial (RCT) to evaluate the clinical and cost-effectiveness of the intervention in improving outcomes for pwMS during transition to SPMS.

PRIMARY OBJECTIVE

The primary objective is to assess the acceptability and credibility of an acceptance-based telephone support intervention provided during the transition to SPMS through a feasibility RCT aimed at increasing physical activity and improving social relationships. This follows NICE guidance towards recommendations for increasing activity in MS and research evidence highlighting the importance of maintaining the psychological wellbeing of patients during transition to SPMS and the importance of social relationships within this.

SECONDARY OBJECTIVES

The secondary objectives are to demonstrate proof of principle of the intervention by gathering information about the process of change between the two treatment arms on self-efficacy, emotional coping, and mood, and to gather feedback, through nested interviews, on the intervention and study procedures.

TRIAL / STUDY DESIGN

TRIAL / STUDY CONFIGURATION

A single centre mixed methods feasibility randomised control trial (fRCT) is to be conducted to assess the feasibility and optimal delivery of the acceptance based support intervention with people recently diagnosed with SPMS. The fRCT will have two groups: (1) Acceptance Based Support + Usual Care (ABS+UC) and (2) Usual Care (UC). Participants will be assessed at Baseline, and then again at 8 and 12 weeks post-randomisation, with participation in the study taking an estimated 4 months. A selection of the participants will then be invited to complete feedback interviews. UC refers to the typical contact made to those recently diagnosed with SPMS by the Neurology service.

Primary endpoint

The primary endpoints in this study relate to the feasibility of proceeding to a future RCT.

1. Acceptability and feasibility of trial procedures
2. Appropriateness of eligibility criteria, baseline and outcome measures, audio recording of sessions and randomisation protocol
3. Success of recruitment strategy
4. Recruitment and retention rates
5. Estimation of sample size needed for a future RCT
6. Completion rates of outcome measures

   Secondary endpoint

   The secondary endpoints are to demonstrate proof of principle of the intervention by gathering information about the process of change between the two treatment arms on self-efficacy, emotional coping, and mood, and to gather feedback, through nested interviews, on the intervention and study procedures.

   RANDOMIZATION AND BLINDING

   Once the decision to include a pwMS is made, they will be randomised to one of two groups in a ratio of 1:1: (1) ABS+UC or (2) UC. Block randomisation of 2, 4, 6 and 8 will be used to ensure parity between groups, and randomly selected block sizes will be used to avoid selection bias. Randomisation will be conducted using an online sealed envelope service (www.sealedenvelope.com), to generate a priori the random allocation sequence. Trial researchers will access the allocation for each participant by logging in to this remote, secure internet-based randomisation system. Once a participant has consented to the study and completed the baseline measures, the researcher will log into the randomisation system and enter basic demographic information to receive the allocation for that participant. The sequence of treatment allocations will be concealed until interventions have all been assigned and recruitment, data collection, and all the other assessments are complete.

   TRIAL/STUDY MANAGEMENT

   The University of Nottingham (UoN) will act as the Sponsor for the trial. UoN's Standard Operating Procedures (SOPs) will be used to govern the conduct of all aspects of the study. The Sponsor will ensure the trial is run in accordance with our University's SOPs. The trial will be managed and co-ordinated from the Division of Psychiatry and Applied Psychology, School of Medicine, University of Nottingham by the Trial Management Group (TMG), consisting of all of the authors. The trial is funded by the Health Education East Midlands.

   The Trial Management Group (TMG) will meet bi-monthly to ensure milestones are achieved as planned, and will be responsible for the day to day management of the trial. This includes reviewing recruitment, randomisation, retention, data management, adherence to protocol, patient safety, delivery and fidelity of the intervention, data quality and timescales. The TMG will consist of all authors; the Chief Investigator (RdN), Trial Manager (CM), Research Clinical Psychologist (NM), Research Fellow (GT), and Field Supervisor (NE). The Trial Manager (referred to from here as TM) will contact other co-authors for support should issues arise between TMG meetings.

   The CI has overall responsibility for the study and shall oversee all study management.

   The data custodian will be the CI.

   Recruitment

   Participants will be identified within 6 months of receiving a diagnosis of SPMS at the Neurology Clinic at Queens Medical Centre (QMC, Nottingham) and will be told about the study by their treating Neurologist or MS Nurse Specialist. If the potential participant is interested in finding out more about the study, the treating clinician will gain their written consent to contact which will be held in the study files, and their contact details will be passed to the TM. The TM will make telephone contact within one week to confirm their willingness to participate. If they are not interested, the pwMS will be thanked for their time and excluded from the study. No further contact will be made by the TM and their details will be permanently deleted.

   Should the pwMS be interested in participating, the TM will send them an 'Information for Participant' sheet and a copy of the consent form in the post or by email (based on participant preference), and they will be informed that the TM will contact them over the telephone in one week, which should give the material time to arrive and be read. This call will enable the TM to enquire whether they have received the information, allow them to explain the study in more detail, and answer any questions the interested participant has about the study. If they are no longer interested, the person will be thanked for their time and excluded from the study.

   If the participant is still interested in participating, then a pack of outcome measures will be posted to them, and they will be asked to complete these once they arrive. The participant will be instructed to sign and return the consent form, and outcome measures using the pre-paid envelope provided. Completing the consent forms and outcome measures can also be done online, based on participant preference, which may help those participants who are less readily able to travel. Once the consent form, and outcome measures have been returned and the inclusion criteria have been determined to be met, the person will be included in the study.

   Twelve participants, six from each study arm, will be invited to take part in qualitative interviews by the TM following their involvement in the study. These participants will be telephoned to enquire about their interest, and if they would be interested, will be posted or emailed (depending on preference) a Participant Information Sheet (PIS) and a consent form.

   It will be explained to the potential participant that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time but attempts will be made to avoid this occurrence. In the event of their withdrawal it will be explained that their data collected so far cannot be erased and the investigators will seek consent to use the data in the final analyses where appropriate.

   Removal of participants from therapy or assessments/Participant Withdrawal

   Participants will be informed through the PIS and consent form that they are free to withdraw from the study at any time without it affecting their normal care or legal rights. The TM will attempt to replace those who withdraw from the study before randomisation however since this is a feasibility study, participants who withdraw from the study after randomization will not be replaced, but withdrawal rates and reasons will be recorded (if the participants choose to give them). If a participant indicates a wish to withdraw from the intervention, the investigators will enquire whether they will consider completing the follow-up assessments.

   Participants may be withdrawn from the trial either at their own request or at the discretion of the TMG after discussion. If the participant requests to withdraw, efforts will be made to contact the participant over the telephone or other preferred method to understand and respond to their concerns. If participants continue to express they want to withdraw, or do not respond, then they will be considered to have withdrawn. The participants will be made aware that this will not affect their future care. Participants will be made aware (via the PIS and consent form) that should they withdraw the data collected to date cannot be erased and may still be used in the final analysis.

   The TMG may remove a participant from the study where significant disease progression makes aspects of the study impossible. e.g. loss of communication.

   Withdrawal from the Acceptance Based Support programme is not considered a safety issue for participants.

   Informed consent

   All participants will provide written informed consent. The Consent Form will be signed and dated by the participant before they enter the trial. The TM will explain the details of the trial and provide a PIS, ensuring that the participant has enough time to consider participating or not. The TM will answer any questions that the participant has concerning study participation. Informed consent will be collected from each participant: one copy of this will be kept by the participant, one will be kept by the TM. Informed consent will be gathered through one of the following routes before they undergo any interventions, this includes postal or online consent.

   Postal: Two copies of the Consent Forms will be posted to participants, who will be requested to sign and date them. The TM will be available to discuss the information sheet and consent form over the telephone with the participants. Once participants sign the Consent Forms and complete the baseline questionnaires, they will return one consent form and the questionnaires to the investigators using the pre-paid envelope provided. They will keep one consent form for their personal records.

   Online: Online informed consent will be created using online survey tools. The 'mandatory response' function of the online survey tool will be used to ensure obtaining consent from the participants. In this way, participants must confirm they have read the information page and each of the ethical statements. Only when they have 'clicked' to confirm each statement will they be able to move forward to the online baseline questionnaires. Should they wish to have a copy of the consent form, they will be able to print the consent page. If they do not have a printing facility, the investigators will print their consent form and send them a hard copy by post.

   For the qualitative interviews, separate informed consent will be collected from the patient participants before undertaking the interviews following the aforementioned procedures. A separate PIS and Consent Form specific to the interviews will be provided.

   Should there be any subsequent amendment to the final protocol, which might affect a participant's participation in the trial, continuing consent will be obtained using an amended Consent Form which will be signed by the participant.

   TRIAL / STUDY TREATMENT AND REGIMEN

   The investigators will test the feasibility and optimal delivery of the acceptance based support intervention with people recently diagnosed with SPMS, by comparing two groups: (1) Acceptance Based Support + Usual Care (ABS+UC) and (2) Usual Care (UC).

   Interventions:

   Acceptance Based Support + Usual Care (ABS+UC)

   The ABS+UC arm will comprise appointments with the TM who will receive training and supervision from an experienced clinical psychologist (the CI). This will take place over a maximum of 6 sessions, with the first being a face to face session (60 minutes) and the remaining delivered over telephone (30 minutes each). The content of the sessions will be an acceptance based psychological support approach to tackling maintenance of physical activity, and social avoidance. This will comprise of resources which teach an Acceptance and Commitment Therapy (ACT) informed approach to wellbeing, and will be tailored to the specific needs of the participant. A "Patient Workbook", developed from previously designed self-help formats for ACT will be given to all patients in the ABS+UC arm of the study. The workbook will be used as a supplement to assist the guidance and support of the therapist and will not be a standalone self-help intervention, following the recommendations of a recent systematic review and a subsequent thesis.

   Usual Care

   In the UC arm, the participant will meet once with the TM face to face to be informed of the group they have been randomised into and encouraged to ask any questions, and will be informed they will be contacted again in 8 and 12 weeks and be asked to complete some more outcome measures.

   An encrypted UoN dictaphone will be used to audiotape a proportion (10%) of the telephone intervention sessions. Audiotaping will take place in a practical way ensuring that different time points of the intervention are captured. Fidelity to the ACT intervention will then be cross-checked through comparing it against existing criteria to ensure integrity to the model as outlined in an assessment manual.

   Baseline and follow-up assessments

   Participants will be assessed before randomisation at baseline. They will also be assessed at 8 and 12 weeks after randomisation for follow up.

   Demographic data and illness data will be collected at baseline, along with a number of outcome measures detailed looking at mood, psychological flexibility, self efficacy etc. The outcome measures will also be collected at follow up.

   Participant Feedback Interviews

   After the final participant has been randomised, up to 12 participants, six from the ABS+UC and six from the UC condition, will be invited to take part in 30-minute, semi-structured interviews about their experience of the study. A separate information sheet and consent form will be completed in relation to the interviews. Participants will be selected for interview through purposive maximum-variation sampling based on demographic and illness data. An interview schedule will be used and applied flexibly. A 12-participant sample is a manageable number for a study of this size.

   The interviews will be conducted by a trainee clinical psychologist researcher (under supervision from a qualified clinical psychologist with an expertise in qualitative methods) independent of the trial team who will explore the pwMS's experience of receiving each condition, (i.e. what they found helpful or unhelpful, the content and delivery of the intervention). Audio recording will be taken for all interviews and will be transcribed verbatim. An external person/company will be used for transcribing the interviews. A confidentiality agreement will be in place before transferring the interview data to the external company. The transcribed data will be analysed using a framework approach which is a hierarchical, matrix-based method developed for applied qualitative research. Using this approach is appropriate as our goals are clearly defined at the onset (i.e. to support the development of a future definitive trial).

   STATISTICS

   Methods

   Qualitative Analysis

   The feedback interviews will be transcribed by an external (GDPR compliant, and approved by University of Nottingham) transcription service, and analysed by the TM using NVivo data analysis software. A five step Framework Analysis approach will then be taken. This approach involves use of a thematic framework a priori which helps to guide the content of the interviews, which is appropriate for this study as the investigators have clearly defined goals from the outset (i.e. to examine the feasibility of a future RCT trial).

   In Framework Analysis, the data will be mapped onto a constructed thematic framework. After mapping all the data, a matrix will be generated in which the data will be charted to summarise each main theme. This matrix will then be used in the interpretation of the data - in addition to the notes made during the coding process. To ensure rigour and credibility of the findings, the generated matrix will be reviewed by another researcher and the quotations for their relevance to the themes will be checked. Disagreements will be resolved by discussion in the TMG.

   Quantitative Analysis

   As a feasibility trial, the main analysis will be descriptive and focus on confidence interval estimation and not formal hypothesis testing. Descriptive statistics will be used to describe outcomes and to inform power and sample size calculations for a future trial. Rates of consent, recruitment and follow-up by randomised groups will be reported. Based on the characteristics of the data, appropriate parametric and non-parametric statistics will be used to describe trends.

   SPSS for Windows will be utilised for the analysis of outcome measures, illness and demographic data, and feasibility measures (e.g. number of missed appointments). Frequencies and percentages of missed and rescheduled support calls, attrition rates and adherence to outcome measures will be gathered. In addition, analysis of variance (ANOVA) will be used to explore outcome data at different time-points, to allow for calculation of effect sizes to help ascertain sample size predictions for a future RCT. Regression will be used to help the investigators predict the likelihood of change, using initial HADS scores, illness, and demographic factors as variables.

   Sample size and justification

   The recruitment target is to randomise 40 pwMS, based on recommended sample sizes between 24 and 50 for feasibility RCTs. Recruiting 15 participants or above per study condition is considered acceptable to obtain a reasonable sample size estimate for pilot trial studies, and recent similar research of an 8-session telephone study comparing CBT to supportive listening showed a consistent attrition rate across interventions with this population of around 15%. Therefore, a slightly larger target (20 per arm) for 6 sessions will help to prepare for the possibility of a 25% attrition rate, whilst still achieving the 15 participants per arm suggested to evidence a future RCT. An estimation for the recruitment rate is to recruit five participants each month, between March 2019 and October 2019.

   DATA PROTECTION

   All trial staff and investigators will endeavour to protect the rights of the trial's participants to privacy and informed consent, and will adhere to the Data Protection Act, 2018. The CRF will only collect the minimum required information for the purposes of the trial. CRFs will be held securely, in a locked room, or locked cupboard or cabinet. Access to the information will be limited to the trial staff and investigators and relevant regulatory authorities (see above). Computer held data including the trial database will be held securely and password protected. All data will be stored on a secure dedicated web server. Access will be restricted by user identifiers and passwords (encrypted using a one way encryption method).

   For online consent and questionnaires, an online survey tool (e.g. Online Surveys) will be used, which complies fully with the General Data Protection Regulation. The investigators will set up an account dedicated for the AT-SPMS study (only the research team members will have access to this account). All online responses will be collected over encrypted SSL connections and stored on the password-protected AT-SPMS online survey account. The account will be checked by the research team on a weekly basis to export the collected online data to a secure dedicated web server (Access will be restricted by user identifiers and passwords). Once the online data (i.e. stored on the online survey account) is exported to this secure dedicated web server, it will be permanently deleted from the online survey account. Automatic IP collection option would be turned off to maintain the participants anonymity.

   Information about the trial in the participant's medical records / hospital notes will be treated confidentially in the same way as all other confidential medical information.

   Electronic data will be backed up every 24 hours to both local and remote media in encrypted format.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to consent to the trial
2. Have received a diagnosis of SPMS in the last 1 year
3. Are 18 years or over (no upper age limit)
4. Score greater than 7 (indicating clinical severity) on either subscale of the Hospital Anxiety and Depression Subscale (HADS)
5. Able to communicate in English

Exclusion Criteria:

1. Are currently receiving any psychological or cognitive intervention for their mental health (or received this in the last 3 months)
2. Are participating in another concurrent interventional study
3. Have a severe co-morbid psychiatric condition (e.g., dementia), as reported by patients or by the clinical team making the initial approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
The administrative burden of the trial for participants and for investigators, measured through feedback interviews and hours per week necessary to facilitate the trial | 4 months (length of participant journey through the study)
  The administrative burden of the trial, for both the investigators and the participants will be recorded. For the participants, this will be investigated through the feedback interviews. For the investigator, this will be a measure of how many hours it takes per week to facilitate the trial.
The appropriateness of the overall eligibility criteria, such as the total number, and ratio, of participants being included/excluded by each criteria. | 4 months
  The appropriateness of the eligibility criteria will be measured through recording the numbers of eligible participants in the service, to ensure they are not too restrictive/too inclusive when considering the sample needed and the time available. The total number, and ratio, of participants being included/excluded by each criteria will be gathered.
  This will be important for any future trial to estimate the time it would take to recruit using the eligibility criteria.
The ease and success of the randomisation protocol, measured through the amount and frequency of any errors (see description) during the randomisation process. | 4 months
  The ease and success of the randomisation protocol (using Sealed Envelope, SealedEnvelope.com) will be assessed, and any errors or difficulties in useability will be recorded (e.g., being unable to access the randomisation system to randomise a participant promptly, or there being a large disparity between numbers randomised in each group) .
Acceptability of audio recording of sessions: number who accept, decline | 4 months
  The response of participants (number who accept, decline) to being audio recorded to assess fidelity of the therapy will be measured.
Success of recruitment/ recruitment rates | 4 months
  The number of participants identified as eligible for the study (meeting all inclusion criteria) and contacted will be recorded, along with the number who agree to take part.
Retention rates | 4 months
  The number of participants who complete the study procedures, or drop out, and for what reasons, will be recorded.
Completion rates of outcome measures | 4 months
  The type and amount of missing data found on each questionnaire and whether this missing information could be obtained by telephone follow-up will be determined. These data will also indicate any problems of outcome questionnaires being sent by post and the ease of answering these.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) | 4 months
  An anxiety and depression assessment. The minimum score is 0 and the maximum score is 42 (21 for anxiety, 21 for depression). A higher score indicates a greater level of distress.
  The scores from the questionnaires will be used to compute sample-size and power calculations for a future RCT.
Multiple Sclerosis Impact Scale-29 (MSIS-29) (Riazi, Thompson, Lamping, Hobart, & Fitzpatrick, 2001) | 4 months
  A perceived physical and psychological impact of MS assessment. The minimum score is 29 and the maximum score is 145. A higher score indicates a greater impact of multiple scleorosis on the individual.
  The scores from the questionnaires will be used to compute sample-size and power calculations for a future RCT.
Multiple Sclerosis Self-Efficacy Scale (Rigby et al., 2003) | 4 months
  An efficacy (extent to which pwMS feel in control and able to overcome the challenges they are faced with) assessment.
  The minimum score on this measure is 14, the maximum score is 84. Higher scores indicate greater self efficacy.
  The scores from the questionnaires will be used to compute sample-size and power calculations for a future RCT.
EQ-5D-5L (Herdman et al., 2011) | 4 months
  A Health-related Quality of Life (QoL) assessment split into two sections.
  Section 1 assesses: mobility, self care, usual activities, pain/discomfort and anxiety/depression.
  The minimum score is 5, the maximum score is 25. A higher score indicates a lower quality of life.
  Section 2 is a single item rating of a person's "health today" (0-100). Higher scores indicate better health.
  The scores from the questionnaires will be used to compute sample-size and power calculations for a future RCT.
Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT) (Francis, Dawson, & Golijani-Moghaddam, 2016) | 4 months
  A process measure to show proof of principle in Acceptance and Commitment Therapy (ACT).
  It has a minimum score of 0, and a maximum score of 138. A higher score indicates greater psychological flexibility (constituting openness, awareness, activation)
  The scores from the questionnaires will be used to compute sample-size and power calculations for a future RCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Queens Medical Centre, Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data collected will be anonymised. No individuals data will be distributed or identifiable.